CLINICAL TRIAL: NCT01515514
Title: Confocal Endomicroscopy for GI Neoplasia Study
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Bankhead-Coley (Unknown)
Responsible Party: Principal Investigator, Michael Wallace, Primary Investigator, Mayo Clinic
Other Study IDs: 11-006327
Record Dates: First submitted 2012-01-10; First posted 2012-01-24 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Colorectal Polyps
Keywords: polyps; inflammatory bowel disease; associated neoplasia
MeSH Terms: conditions — Polyps; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to enhance probe stabilization using a 4mm clear cap attached to endoscope in comparison to standard "free-hand" image acquisition.

DETAILED DESCRIPTION:
The aim of this study is to optimize and validate in-vivo imaging systems capable of highly accurate, real-time classification of colorectal neoplasia.

ELIGIBILITY:
Inclusion Criteria:

* Those patients undergoing colonoscopy for screening or surveillance of colon polyps will be included in this study.

Exclusion Criteria:

* Patients with known polyposis syndromes, inflammatory bowel disease, allergy to fluorescein, or refusal to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 40 patients with polyps
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Quality of the confocal image | 1 yr
  Quality will be assessed subjectively. Subjective technical quality of each video sequence will be scored by two independent experts.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Wallace, MD,MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States